CLINICAL TRIAL: NCT00295204
Title: Evaluation of a Mobile Cardiac Outpatient Telemetry System (CardioNet) Versus Standard Loop Event Monitor: A Multi-Center Randomized Study
Brief Title: Evaluation of a Mobile Cardiac Outpatient Telemetry System Versus Standard Loop Event Monitor
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cardionet (Industry)
Other Study IDs: 05-002
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2006-08-03 (Estimated); Status verified 2006-02

CONDITIONS: Syncope; Pre-Syncope; Palpitations
Keywords: Syncope; pre-syncope; palpitations
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Comparing the arrhythmia diagnostic yield of MCOT as compared to standard loop event monitors in patients presenting with palpitations, syncope or near syncope occurring less frequently than every 24 hours. Patients randomized and are enrolled for 30 days. Prior testing required: 24 hours of non diagnostic monitoring,

DETAILED DESCRIPTION:
Cardiac monitoring is used for diagnosing patient with symptoms. Holter monitoring or cardiac loop monitoring are the tests most ofter prescribed for patients depending on the frequency of symptoms. If the symptoms occur daily, a Holter may be prescribed, but when the symptoms become less frequent the diagnostic yield of Holter monitoring declines greatly. The current yields are approximately 5-10% depending on the indication. When the Holter is not longer an option for patients with infrequent symptoms a cardiac loop event monitor is prescribed to make a diagnosis. The yields on this monitoring also average approximately 25-35%. We feel that the yield on the Mobile Cardiac Ouptatient Telemetry (MCOT) service proviced by CardioNet is significantly higher due to the fact that every beat is analyzed using an algorithm and that many times the arrhythmia causing the symptoms has ended before the patient is able to press the button on the loop monitor to record the ECG. This study compares the MCOT service with Patients over 18 years of age experiencing syncope, near syncope or palpitations less frequently than daily. Require 24 hours of non-diagnostic ECG monitoring prior to randomization. Patients remain on monitoring for 30 days unless an arrhythmia diagnosis is made. The primary endpoint is confirmation of exclusion of a probable arrhythmic cause of pre-syncope, syncope or palpitations experienced by the subject prior to enrollment in the study. Secondary endpoints include time to diagnosis, time to detection of clinically significant arrhythmias, comparison of non-clinicaly significant arrhythmias, rate of asymptomatic arrhythmias both clinically and non clinically significant and a diagnosis related resource utilization. The study size is 300 subjects.

ELIGIBILITY:
Inclusion Criteria:

* syncope, pre-syncope or palpitations less frequently than every 24 hours Pre-syncope without loss of consciousness defined as transient dizziness, leghtheadedness, unsteadiness or weak spells: syncopal events with or without warning: palpitations Subjects with non-diagnostic 24 hours of monitoring related to symptoms within 45 days of enrollment into study Subject able to understand, assent to , and willing to sign the Informed Consent Form.

Exclusion Criteria:

* Class IV heart failure Post Myocardial infarction less than or equal to 3 months Unstable angina defined as chest pain at rest, new onset of angina, or a change in existing patterns of angina.

Subjects who are candidatees for or have had recent (less than or equal to 3 monthr) heart valve surgery History of sustained ventricualr tachycardia or ventricular fibrillation documented EF 35% or less with complex ectopy defined as PVC's 10 or greater per hour.

Subject is less than 18 years old at the time of signing informed consent. Any condition which may prohibit the completion of or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-04; Study Completion 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Rothman, MD, Principal Investigator — Mainline Arrhythmia and Cardiology Associates
Locations (13):
- United States (13):
  - Medicor Cardiology, PA, Bridgewater, New Jersey
  - Garden State Cardiovascular Associates, Elizabeth, New Jersey
  - Monmouth Cardiology Associates, LLC, Ocean City, New Jersey
  - Cardiovascular Associates of NY, Flushing, New York
  - Abington Medical Specialists, Abington, Pennsylvania
  - Central Bucks Cardiology, Doylestown, Pennsylvania
  - Central Bucks Specialitsts, LTD, Doylestown, Pennsylvania
  - PA Heart and Vascular Group, Jenkintown, Pennsylvania
  - Lancaster Heart and Stroke Foundation, Lancaster, Pennsylvania
  - Southwestern PA Cardiology Associates, Pittsburgh, Pennsylvania
  - Pottstown Medical Specialistsq, Pottstown, Pennsylvania
  - Cardiology Consultants of Phladelphia, Yardley, Pennsylvania
  - Virginia Cardiovascular Specialist, Richmond, Virginia